CLINICAL TRIAL: NCT07136623
Title: Deep Learning for Algorithmic Detection of Pulmonary Hypertension Using a Combined Digital Stethoscope and Three-lead Electrocardiogram
Brief Title: Detecting Pulmonary Hypertension With the Eko CORE 500 Digital Stethoscope
Acronym: EKO-PH
Status: Recruiting | Type: Observational
Sponsor: Eko Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024.4
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pulmnary Hypertension
Keywords: pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Outpatient Echo/RHC Patients: Outpatient Echo/RHC Patients
  Adults (≥18) referred for clinically indicated transthoracic echocardiography (TTE) and/or right heart catheterization (RHC). One study visit (~20 minutes) to obtain ≥4 15-second Eko CORE 500 recordings (phonocardiogram and three-lead electrocardiogram) at standard auscultation sites. No randomization or changes to standard care; investigational algorithm outputs are not used clinically. TTE and/or RHC performed within ±7 days provide reference labels for presence/severity of pulmonary hypertension.
  Interventions: Diagnostic Test: Eko CORE 500 phonocardiogram (PCG) recording; Diagnostic Test: Eko CORE 500 three-lead electrocardiogram (ECG) recording

INTERVENTIONS:
Diagnostic Test: Eko CORE 500 phonocardiogram (PCG) recording — Noninvasive acquisition of heart sound (phonocardiogram, PCG) recordings using the FDA (U.S. Food and Drug Administration)-cleared Eko CORE 500 digital stethoscope. At least four 15-second recordings are collected at standard auscultation sites (aortic, pulmonic, tricuspid, mitral). Recordings are used solely for investigational algorithm development and are not used for diagnostic or clinical decision-making.
  Other Names: Eko CORE 500
Diagnostic Test: Eko CORE 500 three-lead electrocardiogram (ECG) recording — Noninvasive acquisition of three-lead electrocardiogram (ECG) signals using the FDA-cleared Eko CORE 500 digital stethoscope. Recordings are obtained simultaneously with PCG at auscultation sites. Data are used solely for investigational algorithm development and are not intended for diagnostic use.

SUMMARY:
This prospective, observational study will evaluate whether synchronized heart sound (phonocardiogram, PCG) and three-lead electrocardiogram (ECG) recordings (entered as separate interventions in PRS, though collected together in practice) collected with the Eko CORE 500 can help screen for pulmonary hypertension (PH). Adults (≥18 years) undergoing clinically indicated transthoracic echocardiography (TTE) and/or right heart catheterization (RHC) will complete one study visit (~20 minutes). During the visit, study staff will obtain at least four 15-second CORE 500 recordings (aortic, pulmonic, tricuspid, and mitral areas). The clinical echocardiogram (and RHC, if performed) within ±7 days of the recordings will provide reference labels for the presence and severity of PH; de-identified demographic and clinical data may also be abstracted from the medical record.

The primary objective is to develop and validate a software algorithm to detect PH and, where possible, stratify severity using noninvasive PCG+ECG signals. These recordings are investigational data acquisitions for algorithm development only; they are not diagnostic procedures and will not be used for clinical decision-making. Primary performance measures are sensitivity and specificity versus echocardiogram and RHC references. No clinical decisions will be based on the investigational algorithm, and no changes to standard care are required. The study plans to enroll up to ~1,513 participants to obtain approximately 1,375 evaluable datasets across multiple outpatient sites.

DETAILED DESCRIPTION:
This is a prospective, observational, multi-site study to determine whether synchronized heart-sound (phonocardiogram; PCG) and three-lead electrocardiogram (ECG) recordings (entered as separate interventions in PRS, though collected together in practice) collected with the FDA (U.S. Food and Drug Administration)-cleared Eko CORE 500 digital stethoscope can assist in screening for pulmonary hypertension (PH). Adults (≥18 years) referred for clinically indicated transthoracic echocardiography (TTE) and/or right heart catheterization (RHC) will complete a single study visit (~20 minutes). During the visit, trained staff will obtain at least four 15-second CORE 500 recordings from standard auscultation locations (aortic, pulmonic, tricuspid, and mitral).

The clinical TTE (and RHC, if performed) completed within ±7 days of the recordings will provide reference labels for the presence and severity of PH. If available, de-identified results from a clinical 12-lead ECG performed within 30 days of the TTE may also be abstracted for comparison. The primary objective is to develop and validate a software algorithm that detects PH from PCG+ECG signals; secondary objectives include assessing severity stratification and overall diagnostic performance (e.g., sensitivity/specificity, area under the receiver operating characteristic curve [AUC], positive predictive value [PPV], negative predictive value [NPV]), including subgroup analyses to evaluate generalizability. These recordings are investigational data acquisitions for algorithm development and detection research only; they are not diagnostic procedures and will not be used for clinical decision-making.

The study plans to enroll up to ~1,513 participants to obtain approximately 1,375 evaluable datasets (about 1,250 with TTE and 125 with RHC). No clinical decisions will be based on investigational algorithm outputs, and participation does not alter standard care. Key eligibility includes adults able to consent who have a clinical TTE or RHC within the protocol window; exclusions include current hospitalization and limited TTE studies. All study data are de-identified using site-maintained key-coded identification codes (IDs). PCG/ECG recordings are transmitted to a HIPAA (Health Insurance Portability and Accountability Act)-compliant, secure server; de-identified demographics, clinical data (e.g., TTE Doppler measures including TR [tricuspid regurgitation] velocity and estimated pulmonary artery systolic pressure, RHC hemodynamics), and relevant reports/images may be abstracted/uploaded per site procedures.

This minimal-risk study has IRB (Institutional Review Board) approval. No independent data monitoring committee is appointed; safety oversight is provided by site investigators with adverse event reporting per IRB policy. There is no cost to participants; modest compensation (≤$50, site-specific) may be provided. The CORE 500 hardware is FDA-cleared; however, the software algorithm evaluated in this study is investigational (not FDA-cleared). The aim is regulatory readiness for potential future submission without committing to a specific regulatory filing as part of this study.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

Able and willing to provide informed consent.

Clinically indicated transthoracic echocardiogram (TTE) or right heart catheterization (RHC) scheduled/performed within ±7 days of the study recording visit.

Exclusion Criteria:

Unwilling or unable to provide informed consent.

Currently hospitalized at the time of study procedures.

If enrolled via TTE path: limited (non-diagnostic) echocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) receiving outpatient cardiovascular care at participating U.S. centers who are scheduled for, or have recently undergone, clinically indicated transthoracic echocardiography (TTE) and/or right heart catheterization (RHC) within ±7 days of the study visit. Participants are recruited consecutively from clinic and echo/RHC schedules; hospitalized patients are excluded. The population will include individuals with and without pulmonary hypertension across diverse demographics.
Sampling Method: Non-Probability Sample
Enrollment: 1513 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve (AUC) for pulmonary hypertension (PH) detection | Study completion (up to 12 months); reference within ±7 days.
  Description: Area under the receiver operating characteristic (ROC) curve (AUC) of the phonocardiogram (PCG) + electrocardiogram (ECG) algorithm for classifying pulmonary hypertension (PH) vs. non-PH using probability outputs; reference is transthoracic echocardiography (TTE) and/or right heart catheterization (RHC) within ±7 days. 95% confidence intervals (CIs) reported.

SECONDARY OUTCOMES:
Positive and negative predictive values for PH detection | Study completion (up to 12 months); reference within ±7 days.
  Positive predictive value (PPV) and negative predictive value (NPV) at a prespecified operating point; reference is transthoracic echocardiography (TTE) and/or right heart catheterization (RHC) within ±7 days. 95% confidence intervals (CIs) reported.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Troy, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD due to consent limitations and proprietary algorithm development; aggregate results will be shared.

REFERENCES:
- [Background] Maron BA, Choudhary G, Khan UA, Jankowich MD, McChesney H, Ferrazzani SJ, Gaddam S, Sharma S, Opotowsky AR, Bhatt DL, Rocco TP, Aragam JR. Clinical profile and underdiagnosis of pulmonary hypertension in US veteran patients. Circ Heart Fail. 2013 Sep 1;6(5):906-12. doi: 10.1161/CIRCHEARTFAILURE.112.000091. Epub 2013 Jun 27. PMID 23811965
- [Background] Choudhary G, Jankowich M, Wu WC. Elevated pulmonary artery systolic pressure predicts heart failure admissions in African Americans: Jackson Heart Study. Circ Heart Fail. 2014 Jul;7(4):558-64. doi: 10.1161/CIRCHEARTFAILURE.114.001366. Epub 2014 Jun 5. PMID 24902739
- [Background] Strange G, Stewart S, Celermajer DS, Prior D, Scalia GM, Marwick TH, Gabbay E, Ilton M, Joseph M, Codde J, Playford D; NEDA Contributing Sites. Threshold of Pulmonary Hypertension Associated With Increased Mortality. J Am Coll Cardiol. 2019 Jun 4;73(21):2660-2672. doi: 10.1016/j.jacc.2019.03.482. PMID 31146810
- [Background] Assad TR, Maron BA, Robbins IM, Xu M, Huang S, Harrell FE, Farber-Eger EH, Wells QS, Choudhary G, Hemnes AR, Brittain EL. Prognostic Effect and Longitudinal Hemodynamic Assessment of Borderline Pulmonary Hypertension. JAMA Cardiol. 2017 Dec 1;2(12):1361-1368. doi: 10.1001/jamacardio.2017.3882. PMID 29071338
- [Background] Maron BA, Hess E, Maddox TM, Opotowsky AR, Tedford RJ, Lahm T, Joynt KE, Kass DJ, Stephens T, Stanislawski MA, Swenson ER, Goldstein RH, Leopold JA, Zamanian RT, Elwing JM, Plomondon ME, Grunwald GK, Baron AE, Rumsfeld JS, Choudhary G. Association of Borderline Pulmonary Hypertension With Mortality and Hospitalization in a Large Patient Cohort: Insights From the Veterans Affairs Clinical Assessment, Reporting, and Tracking Program. Circulation. 2016 Mar 29;133(13):1240-8. doi: 10.1161/CIRCULATIONAHA.115.020207. Epub 2016 Feb 12. PMID 26873944
- [Background] Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier JF, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Simonneau G. Pulmonary arterial hypertension in France: results from a national registry. Am J Respir Crit Care Med. 2006 May 1;173(9):1023-30. doi: 10.1164/rccm.200510-1668OC. Epub 2006 Feb 2. PMID 16456139
- [Background] Frost A, Badesch D, Gibbs JSR, Gopalan D, Khanna D, Manes A, Oudiz R, Satoh T, Torres F, Torbicki A. Diagnosis of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801904. doi: 10.1183/13993003.01904-2018. Print 2019 Jan. PMID 30545972